CLINICAL TRIAL: NCT04353765
Title: Non - Interventional, Retrospective Study Of Cabozantinib Treatment In Patients With Unresectable, Locally Advanced Or Metastatic Renal Cell Carcinoma Who Progressed After Previous Treatment With Checkpoint Inhibitors
Brief Title: Study Of Cabozantinib Treatment In Patients With Unresectable, Locally Advanced Or Metastatic Renal Cell Carcinoma Who Progressed After Previous Treatment With Checkpoint Inhibitors
Acronym: US NIS Cabo
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: F-FR-60000-066
Record Dates: First submitted 2020-04-17; First posted 2020-04-20 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Locally Advanced or Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- cabozantinib arm
  Interventions: Drug: Cabozantinib monotherapy
- non cabozantinib Tyrosine Kinase Inhibitors (TKI) arm
  Interventions: Drug: All authorized TKI monotherapies in advanced RCC per FDA label in advanced RCC

INTERVENTIONS:
Drug: Cabozantinib monotherapy — Intervention description (FDA Label): kinase inhibitor indicated for the treatment of patients with advanced renal cell carcinoma (RCC).
  Other Names: Cabometyx
  Groups: cabozantinib arm
Drug: All authorized TKI monotherapies in advanced RCC per FDA label in advanced RCC — As per authorized FDA label in advanced RCC
  Groups: non cabozantinib Tyrosine Kinase Inhibitors (TKI) arm

SUMMARY:
To understand the epidemiology, treatment patterns and outcomes of patients with metastatic Renal Cell Carcinoma (mRCC). Data from mRCC patients who received cabozantinib versus non-cabozantinib Tyrosine Kinase Inhibitor (TKI) (a type of targeted cancer drug) immediately after Check Point Inhibitor (CPI) treatment (a type of immunotherapy that blocks proteins that stop the immune system from attacking the cancer cells) in US community oncology practices will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of metastatic Renal Cell Carcinoma (mRCC) during the study period (May 01, 2016 to March 31, 2020);
* Patients who received cabozantinib or non-cabozantinib TKI regimens during identification period (May 01, 2016 to September 30, 2019);
* Patients who received CPIs, as monotherapy, or in combination with a cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitor (e.g. ipilimumab+nivolumab), as the latest treatment for mRCC administrated before cabozantinib or other TKI therapy;
* Patients ≥ 18 years of age as of their index date
* Patients who received care at a US Oncology Network site
* Patients with ≥ 2 visits within the US Oncology Network.

Exclusion Criteria:

* Patients enrolled in a clinical trial at any time during index period
* Patients receiving treatment for another documented primary cancer diagnoses during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US Oncology network
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
6 months Real-World Response Rate | From start of index treatment until 6 months of follow up or end of the treatment or death whichever occurs first

SECONDARY OUTCOMES:
Real-World Overall Response Rate | From start of index treatment until end of the treatment or death whichever occurs first
Overall Survival | From start of index treatment until death or end of the study whichever occurs first
Real-World Duration of Response | From date of index treatment response and the earliest date of progressive disease
Real-World Progression Free Survival | From start of index treatment until the earliest of death, end of study database, or evidence of Progressive Disease
Time to treatment discontinuation | From start of index treatment until treatment discontinuation
Treatment dose reductions | From start of index treatment until treatment discontinuation
  Number of patients who had dose reduction/change as compared to the starting dose during index period
Treatment duration | From start of index treatment until treatment discontinuation
Rate of hospitalisations | From start of index treatment until treatment discontinuation
  Number of patients who had been hospitalized (with reason of hospitalization when available)
Drug discontinuation due to its toxicity | From start of index treatment until treatment discontinuation (through study completion)
  Number of patients discontinuing index regimens due to its toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- McKesson Life Sciences, The Woodlands, Texas, United States